CLINICAL TRIAL: NCT02211755
Title: Phase I Trial of the Combination of Bortezomib and Clofarabine in Adults With Refractory Solid Tumors, Lymphomas, or Myelodysplastic Syndromes
Brief Title: Trial of the Combination of Bortezomib and Clofarabine in Adults With Relapsed Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140161; 14-C-0161
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-08-18

CONDITIONS: Neoplasms; Myelodysplastic Syndromes; Lymphomas
Keywords: Purine Nucleoside Inhibitor; Proteasome Inhibitor; Combination Treatment; Solid Tumors; Hematologic
MeSH Terms: conditions — Neoplasms; Myelodysplastic Syndromes; Lymphoma | interventions — Bortezomib; Clofarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Starting doses are clofarabine at 1 mg/m2 IV on days 1 through 5 of a 21-day cycle, and bortezomib at 0.8 mg/m2 subcutaneously on days 1 and 4 of a 21-day cycle.
  Interventions: Drug: Bortezomib plus Clofarabine

INTERVENTIONS:
Drug: Bortezomib plus Clofarabine — The proteasome inhibitor bortezomib and purine nucleoside metabolic inhibitor clofarabine demonstrated greater than additive activity in combination in preclinical xenograft models

SUMMARY:
Background:

- Researchers want to develop better ways to treat cancer. In this study, they will give people with cancer two drugs. These drugs have been used on their own to treat some blood cell cancers.

Objectives:

- To test the safety and efficacy of the drug combination of bortezomib and clofarabine.

Eligibility:

- Adults age 18 and over with advanced cancer that has progressed after receiving standard treatment or that has no effective therapy.

Design:

* Participants will be screened with medical history, physical exam, and scans to measure their tumors. They will also have heart, blood, and urine tests. All of these may be done by their regular doctors.
* Participants will get the study drugs in 21-day cyles. They will stay at the clinic for week 1 of every cycle, then have 2 weeks off.

<TAB>- Bortezomib will be injected under the skin on days 1 and 4.

<TAB>- Clofarabine will be injected in a vein for days 1-5.

* During cycle 1 only, participants will go to the clinic or their doctor to have a physical exam and blood tests at the start of the second and third week.
* Participants will have clinical evaluations throughout the study, including before receiving treatment and then before the start of each cycle.
* Participants may stay in the study as long as they are tolerating the drugs and their tumor is not getting worse.
* Participants will have follow-up for 30 days after the last dose of study drugs.
* The first part of this study tests the safety of different doses of clofarabine and bortezomib.
* The second part of this study involves a separate group of participants who will undergo mandatory research biopsies to learn more about the effects of clofarabine and bortezomib on cancer cells.

DETAILED DESCRIPTION:
BACKGROUND:

The proteasome inhibitor bortezomib and purine nucleoside metabolic inhibitor clofarabine demonstrated greater than additive activity in combination in preclinical xenograft models, justifying the clinical evaluation of this combination for its antitumor activity

OBJECTIVES:

To establish the safety, tolerability, and maximum tolerated dose (MTD) of bortezomib and clofarabine in patients with refractory solid tumors, lymphomas, or myelodysplastic syndromes (MDS)

To determine the molecular effects of the clofarabine-bortezomib combination on biomarkers of cell death and DNA damage in tumor biopsy tissue

To explore the mechanism of action of the bortezomib and clofarabine combination by examining markers of DNA damage and apoptosis in circulating tumor cells before and after treatment

To characterize the changes in MDS residual disease burden that occur with bortezomib and clofarabine treatment

To examine genomic alterations in circulating tumor DNA (ctDNA) that may be associated with response or resistance to clofarabine-bortezomib combination treatment.

ELIGIBILITY:

* Study participants must have histologically confirmed solid tumors or lymphomas or myelodysplastic syndromes that have progressed on standard therapy known to prolong survival or for which no standard treatment options exist
* Age greater than or equal to 18
* No major surgery, radiation, or chemotherapy within 3 weeks prior to entering the study
* Adequate organ function

STUDY DESIGN:

* This is an open-label Phase I trial
* The starting dose of clofarabine will be 1 mg/m2 administered intravenously on days 1 through 5 of a 21-day cycle; bortezomib will be administered at 0.8 mg/m2 subcutaneously on days 1 and 4 of a 21-day cycle.
* Dose escalation will follow a 3+3 design, with dose limiting toxicities defined during cycle 1.
* Dose escalation will proceed in cohorts comprised of two separate groups of patients (one group of patients with solid tumor/lymphoma and one group of patients with MDS), with at least 1 from each group, until hematologic DLT or the second grade 2 hematologic toxicity is observed, at which point, dose escalation will proceed separately for two cohorts: (1) patients with solid tumors/lymphoma and (2) patients with MDS.
* Up to 33 patients will be accrued to a PD expansi n cohort at the MTD to further assess pharmacodynamic endpoints in tumor and blood.

ELIGIBILITY:
-INCLUSION CRITERIA

1. Patients must have:

   * Histologically confirmed solid tumors that have progressed on standard therapy known to prolong survival or for which no standard treatment options exist, or
   * histologically confirmed myelodysplastic syndrome that has progressed on standard therapy or for which no standard treatment options exist. (As of Amendment L, January 2021, the MDS cohort has been closed due to low accrual.)
2. Age greater than or equal to18 years.
3. ECOG performance status less than or equal to 2.
4. Life expectancy of greater than 3 months
5. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count: greater than or equal to 1,500/mcL for solid tumors and lymphomas only
   * Platelets: greater than or equal to 100,000/mcL for solid tumors and lymphomas only
   * Total bilirubin: less than or equal to 1.5 X institutional ULN (<=3 x upper limit of normal in the presence of documented Gilbert's syndrome or liver metastases at baseline)
   * AST(SGOT)/ALT(SGPT): less than or equal to 3 X institutional upper limit of normal

   OR

   less than 5 X institutional upper limit of normal for

   -creatinine: ess than or equal to 1.5 X institutional ULN

   OR

   creatinine clearance greater than or equal to 60 mL/min/1.73 m2 for patients with creatinine levels >1.5 mg/dL
6. Bortezomib and clofarabine have both been assigned to pregnancy category D by the FDA. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for at least 3 months after dosing with study drugs ceases. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of study drug administration.
7. Patients must have completed any chemotherapy, radiation therapy, or biologic therapy >= 3 weeks (or >= 5 half-lives, whichever is shorter) prior to entering the study. Patients must be >= 2 weeks since any prior administration of a study drug in a Phase 0 or equivalent study and be >= 1 week from palliative radiation therapy (patients on study may be eligible for palliative radiotherapy to non-targeted lesions after 2 cycles of therapy at the PI s discretion). Patients must have recovered to eligibility levels from prior toxicity or adverse events. Treatment with bisphosphonates is permitted.
8. For patients enrolled on the expansion cohort, patients must have tumor amenable to biopsy (excisional or incision biopsies of skin or H & N lesions under visualization) and willingness to undergo tumor biopsies.

EXCLUSION CRITERIA

1. Sensory/motor neuropathy >= Grade 2
2. QTc interval (Fridericia formula) > 450 msec for men or > 470 msec for women at study entry; history of congenital long QT syndrome
3. Patients who are receiving any other investigational agents.
4. Patients with active brain metastases, CNS disease, or carcinomatous meningitis are excluded from this clinical trial. Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no

   evidence of progression.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs. Patients who have previously received either clofarabine or bortezomib will be excluded as this may affect accurate determination of the MTD.
6. Uncontrolled intercurrent illness including, but not limited to, serious untreated infection, symptomatic respiratory failure/congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study because bortezomib and clofarabine have been assigned to pregnancy category D by the FDA. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued prior to the first dose of study drug and women should refrain from nursing throughout the treatment period and for 3 months following the last dose of study drug.
8. HIV-positive patients on combination antiretroviral therapy are ineligible because of possible pharmacokinetic interactions with study drugs.
9. Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Safety and MTD | Cycle 1 (21 days)
  To establish the safety, tolerability, and maximum tolerated dose (MTD) of bortezomib and clofarabine in patients with refractory solid tumors or lymphomas or myelodysplastic syndromes

SECONDARY OUTCOMES:
Biomarkers of DNA damage and apoptosis in circulating tumor cells | Baseline, cycle 1 day 1, and cycle 2 day 1
  To determine the effects of the clofarabine-bortezomib combination on biomarkers of DNA damage and apoptosis in circulating tumor cells
Biomarkers of cell death and DNA damage in tumor biopsy tissue | Baseline, cycle 1 day 1, and cycle 2 day 4/day 5
  To determine the effects of the clofarabine-bortezomib combination on biomarkers of cell death and DNA damage in tumor biopsy tissue

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Duechler M, Linke A, Cebula B, Shehata M, Schwarzmeier JD, Robak T, Smolewski P. In vitro cytotoxic effect of proteasome inhibitor bortezomib in combination with purine nucleoside analogues on chronic lymphocytic leukaemia cells. Eur J Haematol. 2005 May;74(5):407-17. doi: 10.1111/j.1600-0609.2004.00406.x. PMID 15813915
- [Background] Kummar S, Chen HX, Wright J, Holbeck S, Millin MD, Tomaszewski J, Zweibel J, Collins J, Doroshow JH. Utilizing targeted cancer therapeutic agents in combination: novel approaches and urgent requirements. Nat Rev Drug Discov. 2010 Nov;9(11):843-56. doi: 10.1038/nrd3216. Epub 2010 Oct 29. PMID 21031001
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0161.html